CLINICAL TRIAL: NCT06748638
Title: Clinical Study on the Application of Lactulose Combined with Linaclotide in Bowel Preparation for Colonoscopy
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Haifeng Lan (Other)
Responsible Party: Sponsor-Investigator, Haifeng Lan, graduate student, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DZQH-KYLL-24-35
Record Dates: First submitted 2024-12-13; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Lactulose; Bowel Preparation
Keywords: Lactulose; Linaclotide; bowel preparation; colonoscope
MeSH Terms: interventions — Lactulose; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lactulose group ( group 1) (Experimental): lactulose oral solution, Duphalac, 15ml/ bag, 6 bags/box
  Interventions: Drug: Lactulose
- Lactulose + linaclotide group（group 2） (Experimental): Lactulose+ linaclotide 290μg (linaclotide capsule, Lingzeshu, 290ug/ capsule, 7 capsules/box) :
  Interventions: Drug: Lactulose+ linaclotide
- 3L PEG group（group 3） (Experimental): Polyethylene Glycol （PEG）：Heshuang, 137.15g/ bag ，
  Interventions: Drug: polyethylene glycol (PEG)

INTERVENTIONS:
Drug: Lactulose — At 20:00 the night before the examination, pour 2 boxes of lactilose into a cup, add 1000ml of water and drink it; 4 to 6 hours before the examination, dissolve the third box of lactulose into 1000ml water, and drink it; Until pale yellow or clear dung water is drawn.
  Arms: Lactulose group ( group 1)
Drug: Lactulose+ linaclotide — 1 capsule of linalotide (290ug) taken orally half an hour before meal at 12:00 noon on the previous day， and two doses were taken after 20:00 according to the above Lactulose-taking method.
  Arms: Lactulose + linaclotide group（group 2）
Drug: polyethylene glycol (PEG) — a bag of PEG was dissolved into 1L at 20:00 1d before the examination, and was drunk at a constant rate within 2h; 4 to 6 hours before the inspection, dissolve the second bag of PEG into 2L water and drink it.
  Arms: 3L PEG group（group 3）

SUMMARY:
This is a single-center, single-blind, randomized controlled clinical study. Participants meeting the inclusion criteria were randomly assigned to lactulose + linaclotide group, lactulose group, and PEG group in equal proportion.

In this study, the effectiveness, tolerability, adverse reactions and prognosis of three intestinal preparation regimens: lactulose -linalotide group, lactulose group and PEG group were compared by evaluating the intestinal cleanliness rate (BBPS score) of patients and quantitative analysis of intestinal bubble under colonoscopy, with a view to improving the intestinal cleanliness rate of colonoscopy subjects.

DETAILED DESCRIPTION:
1. Research program design This study was designed as a single-center, single-blind, randomized controlled clinical study.
2. Entry criteria Patients aged ≥18 years and ≤80 years who need intestinal preparation before colonoscopy.
3. Study sample size In this study, PASS 15 software was used to estimate the sample size. According to previous research data, the intestinal cleanliness rates of lactulose group (experimental group 1), lactulose + linalotide group (experimental group 2) and PEG group (control group) were set to be 86%, 90% and 69.36%, respectively, and the differences between the two experimental groups and the control group were mainly compared in this study. The bilateral test level for both tests was set as α=0.025, and the degree of assurance was 80%, which was allocated in an equal ratio of 1:1:1. Considering that there may be a 20% shedding rate, 148 patients were planned to be included in each group, and a total of 444 patients were to be included.
4. Number of cases The total number of cases was 444, 148 in each group.
5. Case selection 1) Inclusion criteria:

   ① Sign a written informed consent; Age 18-80 years old, gender is not limited; (3) The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale; (4) Non-lactating pregnant women and no pregnancy plan during the test;
   * Do not participate in any clinical trials for 3 months before and during the trial; 2) Exclusion criteria:

     ①Presence of any contraindications to colonoscopy (gastrointestinal obstruction or perforation, severe acute inflammatory bowel disease, toxic megacolon, severe heart failure, renal failure, or liver failure, etc.)

     ② Galactosemia patients;

     ③Pregnancy or lactation;

     ④ Allergic to intestinal preparation drugs;
   * Termination of the experiment for any other reason.
6. Observation index

<!-- -->

1. Main outcome measures: Patients' intestinal cleanliness rate (BBPS score)
2. Secondary outcome measures

   * The number of bubbles in the colonoscopy cavity;

     * polyp detection rate (PDR) and Adenoma detection rate (ADR);

       * Subjects' satisfaction;

         * subject tolerance; (5) Intestinal preparation completion rate;

           * Amount of exercise during intestinal preparation;

             * Colonoscopy operation time;

               * Incidence of adverse reactions; ⑨ Whether to have a colonoscopy for the first time;

                 ⑩ The main indications of colonoscopy;

                 ⑪ Willingness to conduct intestinal preparation;

                 ⑫ Sleep quality. 7.Preparation before treatment:

                 1 or 3 days before colonoscopy, all the three groups were forbidden to eat high-fiber vegetables, dragon fruit and other seeded fruits, and should mainly eat low-fiber and low-residue foods, and eat dinner before 18:00, and then fast; Check for semi-liquid or liquid food the night before, and check for fasting and no drinking on the day.

                 8.Post-treatment: To replace fluid loss during the examination, the patient then drinks an adequate amount of fluid to maintain adequate hydration. Seek medical attention if severe or persistent diarrhea occurs.

                 9.Security assessment: The main adverse reactions were recorded as nausea, vomiting, abdominal distension and abdominal pain.

ELIGIBILITY:
Inclusion Criteria:Participants must meet all of the following criteria to enter the trial.

1. Signed written informed consent;
2. Age 18-80 years old, gender is not limited;
3. The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale;
4. Non-lactating pregnant women and no pregnancy plan during the test;
5. Do not participate in any clinical trials for 3 months before and during the trial;

Exclusion Criteria: Subjects must exclude all of the following conditions to enter the study.

1. Presence of any contraindications to colonoscopy (gastrointestinal obstruction or perforation, severe acute inflammatory bowel disease, toxic megacolon, severe heart failure, renal failure, or liver failure, etc.)
2. Patients with galactosemia;
3. Pregnancy or lactation;
4. Allergic to intestinal preparation drugs;
5. Termination of the experiment for any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation quality | 1 day of scheduled colonoscopy
  The proportion of subjects with an overall Boston score ≥6 and a colon score ≥2 for each segment was considered valid.
  The Boston bowel preparation scale (BBPS) can be used to evaluate indicators such as the volume, shape and mucosal clarity of stool and fluid in the bowel. The scoring criteria are as follows: 0 score: uncleared stool in the colon with indistinct mucosa, most commonly in the stage without bowel preparation; 1: Part of the intestinal mucosa was clearly displayed, while the other part of the mucosa was not clearly displayed due to feces and opaque liquid residues; 2 points: There is a small amount of stool and opaque liquid remaining in the colon; 3 points: All mucous membranes are clearly displayed, and no stool or opaque fluid remains in the colon. Rating description:
  * The colon score of each segment was 0~3, and the total score was 0~9. ② The colon score of each segment was ≥2 points, indicating adequate intestinal preparation; ③ The total score of 6 and the score o

CONTACTS AND LOCATIONS:
Overall Officials: Ji Xuan, Study Director — Jinling Hospital, China
Locations (1):
- Jinling Hospital, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No